CLINICAL TRIAL: NCT06860165
Title: Validation of EmoDTx as a Digital Endpoint for Mood Monitoring in Adult Patients With Unipolar Depression: An Observational Study Against Standard Depression Assessment Questionnaires
Brief Title: Validation of EmoDTx as a Digital Endpoint for Mood Monitoring in Adult Patients Suffering From Unipolar Depression
Acronym: EMC2FR
Status: Recruiting | Type: Observational
Sponsor: Emobot (Industry)
Collaborators: Nîmes University Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: EMC2FR; 2024-A02120-47 (Other: ANSM)
Record Dates: First submitted 2025-02-11; First posted 2025-03-05 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Unipolar Depression; Major Depressive Disorder (MDD); Depression
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to validate the EmoDTx as a digital tool for mood monitoring in adult patients with unipolar depression. The study is prospective, multicenter, and observational, with a single-arm approach. The device studied, EmoDTx, is a mood-monitoring application that analyzes patients' facial expressions to assess their emotional state. The study aims to compare mood scores obtained via EmoDTx with those of standard depression questionnaires (MADRS, PHQ-9, BDI-II, HAMD-17, QIDS-SR16). It will also provide information on how patients feel about the use of passive monitoring software (without the active involvement of the patient) and how the feedback sent to patients can help in their care.

Participants who agree to take part in the study, during a selection visit, will be able to:

1. Install the software on a digital interface (smartphone, computer, etc.) and activate or deactivate it whenever they wish during the 8-week follow-up period.
2. Attend scheduled appointments at the center (a first appointment, then a second 4 weeks later, and a final at 8 weeks) to complete a series of questionnaires, be questioned by the doctor, and fill in other questionnaires on their own.
3. At home, answer questionnaires independently, 2 weeks and 6 weeks after the first appointment.
4. The application's feedback will be deactivated during the first 4 weeks and then reactivated during the final 4 weeks.
5. In parallel, an ancillary study will be conducted on 16 patients enrolled in EMC2FR who accepted and performed the video recording of their structured clinical interview following SCID-5-CV at baseline and 4 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Outpatients diagnosed with mild to severe unipolar disorder
2. Age ≥ 18 years old
3. Patients willing and able to participate (i.e willing to use the EmoDTx App and having the necessary technical equipment to use it)
4. Patients who read, write and understand French
5. Patients having signed the Patient Informed Consent

Exclusion criteria:

1. Patients hospitalized
2. Patients taking more than 75% of the maximal recommended daily dose of benzodiazepines
3. Patients taking more than 75% of the maximal recommended daily dose of antipsychotics
4. Patients taking more than 75% of the maximal recommended daily dose of neuroleptics
5. Patients who did not respond to 10 different pharmacological treatments
6. Patients who attempted suicide within the previous last 6 months and presenting with suicidal ideations
7. Patient presenting with bipolar disorders
8. Patients with a contra-indication to the device under evaluation:

   * Severe depression requiring hospitalization
   * Schizophrenic disorders according to DSM 5 classification
   * Major neurocognitive disorders according to DSM 5 classification
   * Illiteracy
   * Subject hospitalized in a healthcare or social institution for reasons other than biomedical research or is deprived of freedom by administrative or judicial decision or is placed under guardianship
9. Patients unable to read, write and understand French
10. Patients with no access to a smartphone or a computer with an internet connection
11. Patients who refuse to sign the Patient Informed Consent
12. Patients already participating in another interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from mild to severe unipolar depression
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Change of score EmoDTx | From baseline to 4 weeks
  Absolute difference
Change of score MADRS administrated by an investigator | From baseline to 4 weeks
  Absolute difference

SECONDARY OUTCOMES:
Change of EmoDTx score | Between 2 weeks and 6 weeks
Change of score PHQ-9 self reported | Between 2 weeks and 6 weeks
Change of EmoDTx score | Between Baseline and 4 weeks, between Baseline and 8 weeks and between 4 weeks and 8 weeks
Change of HAMD-17 questionnaire administered by the investigator | Between Baseline and 4 weeks, between Baseline and 8 weeks and between 4 weeks and 8 weeks
Change of EmoDTx score | between Baseline and 4 weeks - between Baseline and 8 weeks - between 4 weeks and 8 weeks
Change of score QIDS- SR16 self administrated | between Baseline and 4 weeks - between Baseline and 8 weeks - between 4 weeks and 8 weeks
Change of score BDI-II self administrated | between Baseline and 4 weeks - between Baseline and 8 weeks - between 4 weeks and 8 weeks
Score EmoDTx | At 4-weeks, at 8 week
Score MADRS administrated by the investigator | At 4-weeks, at 8 week
Score HAMD-17 administrated by the investigator | At 4-weeks, at 8 week
Score PHQ-9 self administrated | At 2-weeks and 6 weeks.
Score QIDS-SR16 self administrated | At 4-weeks and 8 weeks
To evaluate the ability of EmoDTx to predict changes in patient's mood earlier than the standard-of-care questionnaires HAMD-17, within 4 weeks and 8 weeks of follow-up. | Time to detection by EmoDTx of changes to depression severity symptoms within 4 weeks and 8 weeks of follow-up as compared to changes detected by standard-of-care questionnaires HAMD-17 Changes in depression severity
To evaluate the ability of EmoDTx to predict changes in patient's mood earlier than the standard-of-care questionnaires MADRS, within 4 weeks and 8 weeks of follow-up. | Time to detection by EmoDTx of changes to depression severity symptoms within 4 weeks and 8 weeks of follow-up as compared to changes detected by standard-of-care questionnaires MADRS Changes in depression severity
Score EQ-5D-5L | At 4 weeks and 8 weeks
Change of EmoDTx score when feedback is deactivated | From baseline to 4 weeks
Change of EmoDTx score when feedback is activated | From 4 weeks to 8 weeks
Acceptability of medical device questionnaire | A baseline and 8 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Cabinet médical Sikorav - Chitic - Roux-Pertus, Changé, France
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No